CLINICAL TRIAL: NCT02388503
Title: The Effect of a Natural Extract on the Post-prandial Blood Glucose Response After Bread Consumption: a Dose-response of Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: FDS-NAA-1946
Record Dates: First submitted 2015-02-10; First posted 2015-03-17 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Healthy
Keywords: Blood glucose
MeSH Terms: interventions — Fruit

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Reference (Placebo Comparator): No added fruit extract
  Interventions: Dietary Supplement: no added fruit extract
- Active 1 (Active Comparator): lowest dose of fruit extract
  Interventions: Dietary Supplement: fruit extract
- Active 2 (Active Comparator): low dose of fruit extract
  Interventions: Dietary Supplement: fruit extract
- Active 3 (Active Comparator): medium dose of fruit extract
  Interventions: Dietary Supplement: fruit extract
- Active 4 (Active Comparator): high dose of fruit extract
  Interventions: Dietary Supplement: fruit extract

INTERVENTIONS:
Dietary Supplement: no added fruit extract
  Arms: Reference
Dietary Supplement: fruit extract
  Arms: Active 1
Dietary Supplement: fruit extract
  Arms: Active 2
Dietary Supplement: fruit extract
  Arms: Active 3
Dietary Supplement: fruit extract
  Arms: Active 4

SUMMARY:
This study is designed to identify the minimal effective tested dose of fruit extract consumed with a bread which provides a reduction in venous post-prandial blood glucose compared to a reference bread.

ELIGIBILITY:
Inclusion criteria:

* Body mass index (BMI) ≥ 18.0 and ≤ 30.0 kg/m2.
* Apparently healthy males and females: no medical conditions which might affect the study measurements including diabetes type 1 and type 2, gastrointestinal dysfunction, gastrointestinal surgery and inflammatory diseases.
* Fasting blood glucose value of subjects ≥ 3.4 and ≤ 6.1 mmol/litre (i.e. 62-110 mg/dl) at screening.

Exclusion criteria:

* Use of antibiotics within 3 months before day 1; use of any other medication except paracetamol, within 14 days before day 1.
* Blood donation in the past 3 months and/or during the study.
* Reported intense sporting activities > 10 h/week.
* Consumption of > 14 units (female subjects) and > 21 units (male subjects) alcoholic drinks in a typical week.
* Reported dietary habits: medically prescribed diet, slimming diet, not used to eat 3 meals a day, vegetarian.
* If female, is pregnant (or has been pregnant during the last < 3 months) or will be planning pregnancy during the study period.
* If female, is lactating or has been lactating in the 6 weeks before screening and/or during the study period.
* Dislike, known allergy or intolerance to test products or other food products provided during the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2015-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Positive incremental post-prandial blood glucose area under the curve | 120 minutes

SECONDARY OUTCOMES:
Post-prandial insulin response | 120 minutes
Post-prandial insulin response | 180 minutes
AUC of fruit extract calculated by a non-compartmental model | 180 minutes
AUC of fruit extract calculated by a population model | 180 minutes
Positive incremental post-prandial blood glucose area under the curve | 180 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Charité research organisation, Berlin, Charitéplatz 1, Germany